CLINICAL TRIAL: NCT01827423
Title: Squamous Cell Carcinoma Antigen as a Marker of Sinonasal Inverted Papilloma
Brief Title: Squamous Cell Carcinoma Antigen Analysis at the University Hospital Ostrava
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FNO-ENT-SCCA
Record Dates: First submitted 2013-03-22; First posted 2013-04-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Nasal Polyps; Nasal Diseases; Papilloma
Keywords: squamous cell carcinoma antigen; sinonasal inverted papilloma; clinical marker; hidden reccurence; surgery
MeSH Terms: conditions — Nasal Polyps; Nose Diseases; Papilloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Surgical removal of sinonasal papiloma (Experimental): The study group consisted of patients following a surgical removal of sinonasal papiloma, in which the SCCA blood levels were assessed in pre-defined intervals.
  Interventions: Device: Surgical removal of sinonasal papiloma

INTERVENTIONS:
Device: Surgical removal of sinonasal papiloma — An endoscopic endonasal surgical device is used to remove the sinonasal papilomas in the study subjects.
  Other Names: endoscopic endonasal surgery

SUMMARY:
This prospective study aimed to evaluate the usefulness of squamous cell carcinoma antigen (SCCA) as a clinical marker of sinonasal inverted papilloma (IP). The potential benefit of SCCA in the diagnosis of unilateral nasal pathology and as a marker of hidden recurrence was evaluated as well.

Blood samples from patients with sinonasal IP were examined to determine serum SCCA levels before surgery, the day after surgery, and every 6 months during follow-up. Preoperative and postoperative levels of SCCA were compared.

DETAILED DESCRIPTION:
INTRODUCTION Squamous cell carcinoma antigen (SCCA) is a protein with a strong homology to the family of protease inhibitors known as serpins. SCCAs are cytoplasmic proteins: they are found in normal squamous epithelia, and in elevated levels in the serum of patients with squamous cell carcinomas, especially in cases of uterine cervix carcinoma, lung carcinoma, and head and neck squamous cell carcinoma. SCCA is clinically useful, especially for the staging of uterine cervix carcinoma (risk of lymph node metastasis). It is also a useful marker for monitoring during follow-up and therapy, and increasing SCCA levels may predict carcinoma relapse. Recent studies have shown a close relationship between SCCA and sinonasal inverted papilloma (IP).

IP is a relatively infrequent, benign sinonasal tumour. Careful long-term follow-up after radical surgery is necessary when treating IP, owing to its malignant potential and high recurrence rate. Distinguishing between inflammatory changes and recurrence of IP can sometimes be difficult. The purpose of this study was to determine the benefit of SCCA serum level evaluation in patients with IP.

MATERIAL AND METHODS Study design This prospective study was performed in accordance with the Declaration of Helsinki, the criteria of good clinical practice, and all applicable regulatory requirements. Written informed consent was obtained from all participants before the initiation of any procedure.

Patients with IP treated at the Department of Otolaryngology, Faculty of Medicine, University of Ostrava were included in the study. At least three years of follow-up after surgery was required for inclusion of a patient in the study.

Blood samples from enrolled patients were examined to determine serum SCCA levels before surgery, the day after surgery, and every 6 months during follow-up. Preoperative and postoperative SCCA levels were compared. The changes in SCCA levels during follow-up were evaluated.

Biochemical analysis Serum SCCA levels were assayed using an immunofluorescence assay with monoclonal antibodies (B.R.A.H.M.S SCC KRYPTOR kit, Hennigsdorf, Germany). The normal serum level of SCC antigen is 0-1.5 µg/l.

Statistical analysis Statistical analysis of the correlation between preoperative and postoperative serum SCCA levels was performed using Student's t-test for paired data. Differences with p < 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* at least three-year follow-up following the surgical procedure
* signed Informed Consent

Exclusion Criteria:

* patient lost during follow-up
* patients in critical condition (ASA IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2000-01; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Changes in blood levels of SCCA before and after surgical removal of sinonasal papiloma | 1 week
  The levels of SCCA were assessed before and after the surgical procedure.

SECONDARY OUTCOMES:
Changes in blood levels of SCCA at six months after surgical removal of sinonasal papiloma | 11 years
  The levels of SCCA were assessed at six months after the surgical procedure and every six months during the follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Kominek, doc.MD,PhD,MBA, Study Director — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

REFERENCES:
- [Background] Yasumatsu R, Nakashima T, Kuratomi Y, Hirakawa N, Azuma K, Tomita K, Cataltepe S, Silverman GA, Clayman GL, Komiyama S. Serum squamous cell carcinoma antigen is a useful biologic marker in patients with inverted papillomas of the sinonasal tract. Cancer. 2002 Jan 1;94(1):152-8. doi: 10.1002/cncr.10144. PMID 11815971
- [Background] Fan GK, Imanaka M, Yang B, Takenaka H. Characteristics of nasal inverted papilloma and its malignant transformation: a study of cell proliferation and programmed cell death. Am J Rhinol. 2006 May-Jun;20(3):360-3. doi: 10.2500/ajr.2006.20.2851. PMID 16871944